CLINICAL TRIAL: NCT03738592
Title: Spatial Hearing Perception in Bilateral Cochlear Implant Children
Acronym: SPHERIC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL18_0471; 2018-A02509-46 (Other: ID-RCB)
Record Dates: First submitted 2018-10-08; First posted 2018-11-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cochlear Impant Children
Keywords: spatial hearing perception; cochlear implant; child; virtual reality
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cochlear implant children (Experimental): 18 cochlear implant children wil include in this study
  Interventions: Other: behavioral exploration of spatial hearing performances; Other: The Speech, Spatial and Qualities of Hearing Scale (SSQ) questionnaire (for cochlear implant children and their parents); Other: The Speech, Spatial and Qualities of Hearing Scale (SSQ) questionnaire (for parents of CI children)
- normal hearing children (Other): 18 normal hearing children wil include in this study
  Interventions: Other: behavioral exploration of spatial hearing performances

INTERVENTIONS:
Other: behavioral exploration of spatial hearing performances — Normal hearing children and cochlear implant children will have to localize a sound source in three dimensional space by using a virtual reality system (Neuro immersion platform). The experiment will last thirty minutes.
  For normal hearing children, this experience will be performed at the inclusion visit.
  For cochlear implant children, this experience will be performed 28 days (+/- 2 days) after inclusion.
Other: The Speech, Spatial and Qualities of Hearing Scale (SSQ) questionnaire (for cochlear implant children and their parents) — For cochlear implant children and their parents, a SSQ questionnaire will be given and completed during the first visit (at the inclusion).
  This questionnaire offers a version for parents of children with hearing loss ("SSQ Parents CI") and a version for the children themselves ("SSQ Children CI").
  Arms: cochlear implant children
Other: The Speech, Spatial and Qualities of Hearing Scale (SSQ) questionnaire (for parents of CI children) — The SSQ questionnaire for Parents of CI children is composed of three distinct sections (A, B and C).
  Each section will be filled separately by parents of CI children with one of the study collaborators during 3 telephone calls spaced 1 week apart. Thus, section A will be completed 7 days (+/- 2 days) after inclusion , section B 14 days (+/- 2 days) after inclusion, and section C 21 days (+/- 2 days) after inclusion.
  Arms: cochlear implant children

SUMMARY:
Spatial hearing in cochlear implant (CI) users is a challenging investigation field since no studies have explored yet spatial auditory perception in three-dimensional space (3D). Moreover auditory rehabilitation after cochlear implantation is totally devoted to speech rehabilitation to date.

A novel methodology based on virtual reality and 3D motion capture protocol in an immersive reality system has recently been developed to evaluate and record spatial hearing abilities of norm-hearing (NH) listeners and CI adults in 3D. The results revealed worse sound localization in 3D for CI users compared to NH participants, and interestingly noted that head movements could improve sound localization performances, leading to a possible track for auditory rehabilitation.

The aim of this study is to explore spatial hearing in CI children with the protocol already tested in CI adults. This protocol will be adapted to children over eight years old. Children will have to perform a sound localization task in 3D without any feedback of performances. The knowledge improvement in pediatric sound localization will lead to develop a specific spatial rehabilitation in cochlear implant children.

ELIGIBILITY:
Inclusion Criteria for cochlear implant children:

* Age between 8 and 17 included
* second cochlear implant issued within more than 2 years
* mean speech recognition over 80% with two cochlear implants
* normal visual acuity with or without correction
* abilities to understand experimental instructions
* a consent form signed by parents or guardian
* registered with a social security scheme

Exclusion Criteria for cochlear implant children:

* neurologic or psychiatric trouble
* visual trouble
* bilateral vestibular areflexia

Inclusion Criteria for normal hearing children:

* Age between 8 and 17 included
* normal visual acuity with or without correction
* abilities to understand experimental instructions
* a consent form signed by parents or guardian
* registered with a social security scheme

Exclusion Criteria for normal hearing children:

* neurologic or psychiatric trouble
* visual trouble
* bilateral vestibular areflexia

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
measure of the spatial hearing deficit matching the distance between the hand pointing error and the sound source position in space | thirty minutes
  Data from spatial sound perception will be recorded in three dimensional space (azimuth, elevation, and depth). First, the pointing error will be computed separately for azimuth, elevation, and depth, in terms of constant error (absolute and signed) and variable error. Then, these separate errors will be combined into a cumulative error "D", hence summarizing all three dimensions of space, and taking into account absolute and variable error in one measure.

SECONDARY OUTCOMES:
measure of head and eye movements in three dimensional space with a motion tracking system (virtual reality system including a Head-Mounted display) to evaluate their roles in spatial hearing performances. | thirty minutes
  Head and eye movements will be recorded in three dimensional space with a motion tracking system (virtual reality system including a Head-Mounted display). The cumulative error "D" will be calculated in two different conditions: first, participant's head will be fixed during sound emission and then, head and eyes will be free to move. If the cumulative error "D" significantly decreases when head movements are free, we could say that head movements allow/help improving spatial hearing performances.
impact of age at cochlear implantation on spatial hearing deficit | thirty minutes
  spatial hearing deficit will be correlated to the age at cochlear implantation
change of the pupil diameter during a sound localization task | thirty minutes
  Pupil diameter will be recorded with an eye tracking system during all experiment
correlation between a clinical score (SSQ) and sound localization performances | 28 days
  The SSQ questionnaire is a clinical subjective scale adapted to parents and cochlear implant children. It allows evaluating hearing performances in daily life. The questionnaire is divided into 3 main items (A: speech; B: spatial hearing; C: other qualities of hearing) comprising questions with rating scores out of ten. For example, a zero score corresponds to bad hearing abilities. We will therefore correlate the mean score of all questions out of ten to the cumulative error "D".

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, PUPH, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Centre de Recherche en Neuroscience de Lyon (CRNL), Bron
  - Hôpital Edouard Herriot, Lyon

REFERENCES:
- [Result] Coudert A, Gaveau V, Gatel J, Verdelet G, Salemme R, Farne A, Pavani F, Truy E. Spatial Hearing Difficulties in Reaching Space in Bilateral Cochlear Implant Children Improve With Head Movements. Ear Hear. 2022 Jan/Feb;43(1):192-205. doi: 10.1097/AUD.0000000000001090. PMID 34225320